CLINICAL TRIAL: NCT05337410
Title: YES: Innovative Discussion for Engagement, Achievement, and Service
Acronym: YES-IDEAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Marc A. Zimmerman, Marshall H Becker Collegiate Professor of Public Health, Center Director, Institute of Firearm Research, Professor of Health Behavior and Health Education, School of Public Health and Professor of Psychology, College of Literature, Science, and the Arts, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00190523; R01MD015024 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-04-20 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Violence Prevention

STUDY DESIGN:
Intervention Model Description: Students enrolled in the YES IDEAS program comprise the treatment group. Students enrolled in other after-school programs (not YES IDEAS) comprise the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YES IDEAS (Experimental): Students participate in the YES IDEAS program.
  Interventions: Behavioral: YES IDEAS
- Control (No Intervention): Students participate in the regular after-school programming.

INTERVENTIONS:
Behavioral: YES IDEAS — YES IDEAS is an adapted version of the evidence based YES (Youth Empowerment Solutions) program. Through the YES program, youth design and implement their own projects to help improve their own communities. The adapted YES IDEAS curriculum empowers youth from various backgrounds to address bullying and promote positive behaviors as a way to reduce violent behavior. Over the course of the program, youth carry out a community change project aimed at promoting non-violence in their community.
  Other Names: YES: Innovative Discussion for Engagement, Achievement, and Service (YES-IDEAS)
  Arms: YES IDEAS

SUMMARY:
The purpose of this study is to evaluate the efficacy of YES-IDEAS (YES: Innovative Discussion for Engagement, Achievement, and Service)compared to regular after school programming in increasing youth empowerment, promoting positive behaviors, and decreasing youth violence.

Through the evidence-based YES (Youth Empowerment Solutions) program, youth design and implement projects to help improve their communities. In the current study, investigators adapted the existing YES curriculum to empower youth from diverse backgrounds to reduce violent behavior. The adapted curriculum, YES-IDEAS, focus on middle school students.

The investigators test the effects of YES-IDEAS curriculum on youths' sense of empowerment, attitudes, and violent behavior. They designed the study to be a group-randomized trial in after-school programs across multiple middle schools in south-east Michigan, but issues that arose due to the COVID-19 pandemic and other practical issues with the schools we modified the design to be a matched control group design at the school level. Matching variables included size, geographic locations, race/ethnicity, free/reduced lunch status. Dose-response and sustainability of YES-IDEAS effects are also examined.

DETAILED DESCRIPTION:
Youth violence is a significant public health concern, as over 20% report being in a fight, 19% reported bullying someone, and 16% reported weapon carriage. Violent victimization among youth includes mental health sequelae in addition to the physical injury caused by violent behavior.

Positive development can be achieved by engaging youth in community improvement activities designed to empower them to avoid risky behaviors. Building on prior research and guided by previous studies of empowerment processes, the investigators developed an afterschool violence prevention program for middle-school students called Youth Empowerment Solutions (YES) for Peaceful Communities. Prior studies have described how YES engages youth in assessing neighborhood assets and liabilities for violence prevention and designing and implementing neighborhood or school projects to reduce violence. Results from prior YES evaluations found the YES program reduced violent behavior and increased positive behaviors in a comparison group design through the process of empowering youth to think critically about their community, develop plans for change, and implement their plans (i.e., program effects were mediated through empowered outcomes).

The existing YES curriculum was adapted to empower youth from various backgrounds to address to address bullying and promote positive behaviors as a way to reduce violent behavior. YES for Engaging Youth for Innovative Discussion for Engagement, Achievement and Service (YES-IDEAS) will focus on middle school students because this is a developmental period when independence from parents begins, their own ideas about peer relationships are formative, and when bullying behavior is at its peak. Empowering children to address violence at this critical developmental period may enable them to resist negative attitudes and behaviors. Working with an advisory board of experts and youth, we will develop and integrate lessons that address these behaviors into the existing YES curriculum.

The study includes two phases: 1) adapting YES and 2) testing YES IDEAS effects. Phase 1 included piloting and evaluating curriculum revisions through testing new modules and obtaining feedback from youth and teachers. Phase 2 tests the effects of YES IDEAS using a matched control trial in after-school programs across multiple middle schools across south-east Michigan. The investigators examine the effects of the curriculum on individual youths' sense of empowerment, attitudes, and violent behavior. Finally, dose-response and sustainability of YES IDEAS effects are examined.

The Specific Aims are:

AIM 1: adapt the YES curriculum to integrate several modules that address youth violence and study the adaptation and implementation process for the new curriculum for middle school students.

AIM 2: Test the efficacy of the YES-IDEAS curriculum in a matched control design on empowered outcomes which will mediate the effects of YES-IDEAS on violent attitudes and behavior.

AIM 3: Investigate if empowered outcomes are the mechanism by which the YES-IDEAS curriculum reduces aggressive and violent behavior over time.

AIM 4: study the effects of dose-response over time on the outcomes from AIMS 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in afterschool programs at multiple middle schools in Counties across south-east Michigan
* Students in 6th through 8th grade
* Students who assent

Exclusion Criteria:

* Non-students
* Students who do not assent or whose parents notify us of their refusal

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 512 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Violence Perpetration | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  6 items on a 4 point Likert scale ranging from 1 (never) to 4 (3 or more times) assess the frequency of physical violence perpetration in the past 30 days. A sample item is "In the past 30 days, how often have you hit someone with your fists or beat up someone?" A higher score indicates more instances of violence perpetration in the past 30 days. Items were adapted for the current study from Hurd et al. (2011).
Change in Targeted Aggression | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  5 items on a 6-point Likert Scale ranging from 1 (never) to 6 (5 or more times) measure frequency of aggression targeted toward specific group in the past 30 days. A sample item includes "In the past 30 days, how often have you told lies or spread false rumors about someone because of their race?" Higher scores indicate more instances of targeted aggression perpetration. Items were adapted for the current study from the Multisite Violence Prevention Project (2004) and Brondolo et al. (2005).
Change in Prosocial behaviors | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  3 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) measure students' prosocial behavior. A sample item is "I am kind to other people." Higher scores indicate more prosocial behavior. Items were adapted for the current study from Nielsen et al., 2015.
Change in Bystander behaviors | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  6 items on a 2-point scale from 0 (no) to 1 (yes) assess youths' bystander behaviors. A sample item is "Have you called out someone who says something bad about another race or makes a racial joke?" Higher scores indicate youth engage in more positive bystander behaviors. Items were adapted for the current study from Salmivalli et al., 1996.
Change in Social action for promoting equity | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  3 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) assess students' behaviors related to social action for promoting equity. A sample item is "I ask questions if people aren't being treated fairly." Higher scores mean more social action. Items were developed for the current study.
Change in Self Efficacy for Inclusion, Diversity, Equity, Acceptance, Solidarity | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  5 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) measure youths' beliefs about their abilities to promote inclusion, diversity, equity, acceptance, and solidarity. A sample item is "I can accept all different types of people." Higher scores indicate more self-efficacy. Items were developed for the current study.
Change in Privilege awareness | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  4 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) measure youths' privilege awareness. A sample item is "Not all racial or ethnic groups have the same chance to get ahead in life." Higher scores indicate greater privilege awareness. Items were developed for the current study.
Change in Recognizing strengths in people | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  3 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) assess youths' recognition of strengths in people. A sample item is "Everyone has something to offer." Higher scores indicate more recognition of strengths in people. Items were developed for the current study.
Change in Social connections across diverse groups | Baseline (0 months), End of Program (3 months), 6 months, 9 months, 12 months
  8 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) assess youths' social connections across diverse groups of people. A sample item is: "I can be friends with someone from a different racial group." Higher scores indicate more social connections across diverse groups. Items were developed for the current study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miao TA, Umemoto K, Gonda D, Hishinuma ES. Essential elements for community engagement in evidence-based youth violence prevention. Am J Community Psychol. 2011 Sep;48(1-2):120-32. doi: 10.1007/s10464-010-9418-6. PMID 21203825
- [Background] Zimmerman MA. Psychological empowerment: issues and illustrations. Am J Community Psychol. 1995 Oct;23(5):581-99. doi: 10.1007/BF02506983. PMID 8851341
- [Background] Zimmerman MA, Stewart SE, Morrel-Samuels S, Franzen S, Reischl TM. Youth Empowerment Solutions for Peaceful Communities: combining theory and practice in a community-level violence prevention curriculum. Health Promot Pract. 2011 May;12(3):425-39. doi: 10.1177/1524839909357316. Epub 2010 Nov 8. PMID 21059871
- [Background] Kellett M. Small shoes, big steps! Empowering children as active researchers. Am J Community Psychol. 2010 Sep;46(1-2):195-203. doi: 10.1007/s10464-010-9324-y. PMID 20524150